CLINICAL TRIAL: NCT00019721
Title: Immunization of Patients With Metastatic Melanoma Using MART-1 and GP100 Peptides Modified to Increase Binding to HLA-0201
Brief Title: Vaccine Therapy With or Without Interleukin-2 in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067051; NCI-99-C-0092; NCI-T99-0033; NCT00001808 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-08-07 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2002-08

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — MART-1 Antigen; aldesleukin; incomplete Freund's adjuvant

INTERVENTIONS:
Biological: MART-1 antigen
Biological: aldesleukin
Biological: gp100 antigen
Biological: incomplete Freund's adjuvant

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells. Interleukin-2 may stimulate a person's white blood cells to kill tumor cells. Combining vaccine therapy with interleukin-2 may be an effective treatment for metastatic melanoma.

PURPOSE: Phase II trial to compare the effectiveness of vaccine therapy with or without interleukin-2 in treating patients who have metastatic melanoma that has not responded to previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of gp100:209-217(210M) peptide and MART-1:26-35(27L) peptide administered with or without high-dose interleukin-2 (IL-2) in patients with metastatic melanoma who are HLA-A0201 positive.
* Determine the efficacy of these peptides in patients who cannot receive IL-2.
* Compare the efficacy of IL-2 with or without these peptides in patients who need immediate treatment with IL-2.
* Determine the efficacy of MART-1:26-35(27L) peptide in patients who have received prior gp100 antigen.
* Compare the immunologic response experienced by patients who have received peptide, with or without IL-2, as measured by changes in T-cell precursors from before to after treatment.
* Compare the toxic effects of these regimens in these patients.

OUTLINE: This is a partially randomized study.

Patients are assigned to 1 of 4 treatment groups based on disease status and prior therapy.

* Group A (eligible to receive interleukin-2 (IL-2) but not in immediate need; no prior immunization with gp100 or MART-1 antigen): Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive gp100 and MART-1 peptides emulsified in Montanide ISA-51 (ISA-51) subcutaneously (SC) on day 1. (Arm I closed as of 10/30/02).
  * Arm II: Patients receive both peptides as in arm I on day 1 and high-dose IL-2 IV over 15 minutes every 8 hours on days 2-5 (for up to 12 doses). (Arm II closed as of 10/30/02).
* Group B (ineligible to receive IL-2 due to other debilitating disease): Patients receive treatment as in group A, arm I.
* Group C (need immediate IL-2 therapy due to extensive and rapid progression of disease): Patients receive treatment as in group A, arm II. (Group C closed as of 10/30/02).
* Group D (prior immunization with gp100 antigen): Patients receive modified MART-1:26-35(27L) peptide emulsified in ISA-51 SC on day 1.

Treatment in all groups repeats every 3 weeks for 4 courses. Patients who achieve a minor, mixed, or partial response may receive up to 12 additional courses. Patients who achieve complete response receive 2 additional courses.

Patients are followed at 4-6 weeks.

PROJECTED ACCRUAL: A total of 103 patients (15-25 for group A, arm I; 19-33 for group A, arm II; and 15 each for groups B, C, and D) will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic melanoma that has failed standard therapy
* Measurable disease
* HLA-A0201 positive

PATIENT CHARACTERISTICS:

Age:

* 16 and over

Performance status:

* ECOG 0-2

Life expectancy:

* More than 3 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 90,000/mm^3

Hepatic:

* Bilirubin no greater than 2.0 mg/dL (less than 3.0 mg/dL for patients with Gilbert's syndrome)
* AST/ALT less than 3 times normal
* Hepatitis B surface antigen negative
* No coagulation disorder

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No major cardiovascular disease
* If cardiovascular disease or other debilitating symptoms present, may receive peptide emulsified with Montanide ISA-51 only

Pulmonary:

* No major respiratory disease

Other:

* Not pregnant
* Fertile patients must use effective contraception
* HIV negative
* No active systemic infection
* No autoimmune disease or immunodeficiency disease
* No primary or secondary immunodeficiency

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 3 weeks since prior biologic therapy
* No prior MART-1 antigen immunization

Chemotherapy:

* At least 3 weeks since prior chemotherapy

Endocrine therapy:

* At least 3 weeks since prior endocrine therapy
* No concurrent steroid therapy

Radiotherapy:

* At least 3 weeks since prior radiotherapy

Surgery:

* Prior surgery allowed

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-04; Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Rosenberg, MD, PhD, Study Chair — NCI - Surgery Branch
Locations (1):
- Surgery Branch, Bethesda, Maryland, United States